CLINICAL TRIAL: NCT02555046
Title: Muscle and Cerebral Oxygenation Under Endovascular Aortic Repair (EVAR) of Abdominal Aortic Aneurysm: General Versus Local Anesthesia - an Randomised Controlled Trial Study
Brief Title: Muscle and Cerebral Oxygenation Under EVAR of AAA: GA vs LA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mads Jacob Niemann, Medical Student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2014-161
Record Dates: First submitted 2015-08-11; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia
Keywords: Spectroscopy, Near-Infrared; Endovascular Procedures; Local Anesthesia; General Anesthesia
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Anaesthesia (No Intervention): EVAR-treatment is preformed with the patient in General Anaesthesia
- Local Anaesthesia (Experimental): EVAR-treatment is preformed with the patient in Local Anesthesia
  Interventions: Procedure: Local Anesthesia

INTERVENTIONS:
Procedure: Local Anesthesia — Use of unspecified local anaesthesia (fx lidocain or bupivacaine)
  Arms: Local Anaesthesia

SUMMARY:
The purpose of this study is to determine the effect of General versus Local Anaesthesia on muscle and cerebral oxygenation under EVAR-treatment in a prospective unblinded randomised controlled trail.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Scheduled procedure

Exclusion Criteria:

* allergies for used local anaesthesia
* have had vascular surgery before in the femoral area
* the need for thromboendarterectomy in common femoral artery
* the need for aortouniiliac stent-graft with cross-over bypass
* severe back pain
* expected time of surgery more than 1.5 hour
* cognitive dysfunction making cooperation during procedure impossible
* Femoral amputee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Near-Infrared Spectroscopy-determined Cerebral Oxygenation | participants will be followed for the duration of hospital stay, an expected average of 5 days
Near-Infrared Spectroscopy-determined Muscle oxygenation | participants will be followed for the duration of hospital stay, an expected average of 5 days